CLINICAL TRIAL: NCT03293524
Title: Efficacy and Safety of Bilateral Intravitreal Injection of GS010: A Randomized, Double-Masked, Placebo-Controlled Trial in Subjects Affected With G11778A ND4 Leber Hereditary Optic Neuropathy for Up to One Year
Brief Title: Efficacy & Safety Study of Bilateral IVT Injection of GS010 in LHON Subjects Due to the ND4 Mutation for up to 1 Year
Acronym: REFLECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-LHON-CLIN-05; 2017-002187-40 (EudraCT Number)
Expanded Access: NCT03672968 (No longer available)
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Leber Hereditary Optic Neuropathy
Keywords: Heredity Optic Atrophy; Leber Hereditary Optic Atrophy; Leber Hereditary Optic Neuropathy; LHON; Eye Diseases; Hereditary Eye Diseases; Inherited retinal dystrophies or degeneration; Inborn Genetic Disease; Gene Therapy; Intravitreal Injections; Mitochondrial Disease; AAV2 Vectors; Nervous System Diseases; Neurodegenerative Disease; Heredodegenerative Disorders of the Nervous System; Atrophy; Pathological Conditions, Anatomical; Anesthetics; Central Nervous System Depressants; Physiological Effects of Drugs
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Eye Diseases; Eye Diseases, Hereditary; Genetic Diseases, Inborn; Mitochondrial Diseases; Nervous System Diseases; Neurodegenerative Diseases; Atrophy; Pathological Conditions, Anatomical

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (Experimental): Subjects will be randomized to treatment arm 1 or treatment arm 2 in a 1:1 allocation. Subjects in treatment arm 1 will receive intravitreal GS010 in both eyes.
  Interventions: Genetic: GS010
- Treatment Arm 2 (Placebo Comparator): Subjects will be randomized to treatment arm 1 or treatment arm 2 in a 1:1 allocation. Subjects in treatment arm 2 will receive GS010 in one eye and placebo intravitreal injection in the other eye.
  Interventions: Genetic: GS010; Drug: Placebo

INTERVENTIONS:
Genetic: GS010 — GS010 is a recombinant adeno-associated viral vector serotype 2 (rAAV2/2) containing the wild-type ND4 gene (rAAV2/2-ND4). GS010 will be administrated via intravitreal injection containing 9E10 viral genomes in 90μL balanced salt solution (BSS) as a single baseline intravitreal injection.
  Other Names: Lenadogene nolparvovec
Drug: Placebo — The placebo is a BSS, sterile, apyrogenic solution and used for ocular surgery. The placebo will be administered via intravitreal injection in a volume of 90 μL.
  Arms: Treatment Arm 2

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of GS010, a gene therapy, in improving the retina functional & structural outcomes in subjects with LHON due to the G11778A ND4 mitochondrial mutation when vision loss duration is present up to one year.

DETAILED DESCRIPTION:
GS-LHON-CLIN-05 is a Phase III, global, multi-center randomized, double-masked for the primary analysis, placebo-controlled, clinical study. As LHON is a neurodegenerative disease, the goal is to administer GS010 as soon as possible upon confirmation of the LHON diagnosis and the causative mutation.

ELIGIBILITY:
Main Selection Criteria:

* Age 15 years or older on the date of signed informed consent.
* Clinically manifested vision loss due to ND4 LHON, to any extent, in at least one eye.
* Vision loss duration of ≤ 365 days (i.e. ≤ 1 year) in each affected eye at Inclusion Visit (Visit 2).

Main Non-Selection Criteria:

* Contraindication to intravitreal injection in any eye.
* Subjects refusing to discontinue idebenone.
* Previous vitrectomy in either eye.
* Narrow angle in any eye contra-indicating pupillary dilation.
* Presence of known/documented mutations, other than the G11778A ND4 LHON-causing mutation, which are known to cause pathology of the optic nerve, retina or afferent visual system.
* History of recurrent uveitis (idiopathic or immune-related) or active ocular inflammation.

Main Inclusion Criteria:

* Vision loss duration of ≤ 365 days (i.e. ≤ 1 year) in each affected eye at Inclusion Visit (Visit 2).
* Each eye of the subject must maintain at least Hand Motion (HM) visual acuity, as defined by the study's SOP for visual acuity testing.
* Documented results of genotyping showing the presence of the G11778A mutation in the ND4 gene and the absence of the other primary LHON-associated mutations (ND1 or ND6) in the subject's mitochondrial DNA.

Main Exclusion Criteria:

* Light Perception (LP) or No Light Perception (NLP) visual acuity in any eye, as defined by the study's standard operating procedure (SOP) for visual acuity testing.
* Presence of active infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye.
* Presence of alcoholism, alcohol dependence, or alcohol or drug abuse (excluding nicotine).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) reported using Log of the Minimal Angle of Resolution (LogMAR) - 1 year | at 1.5 Year post baseline treatment
  The primary efficacy endpoint will be the change from baseline (Visit 2) BCVA reported with LogMAR at 1.5 years post-treatment in second affected/not yet affected eyes of ND4 LHON subjects with vision loss up to one year. The change from baseline (Visit 2) in second affected/not yet affected eyes receiving GS010 and placebo will be the primary response of interest. LogMAR BCVA will be used to represent BCVA.

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) reported with LogMAR - 2 years | at 1.5-Year and 2-Years post baseline treatment
  Change from baseline in LogMAR BCVA at each timepoint of the follow-up period and at 2 years post-treatment.
Responder Analysis | at 1.5-Year and 2-Years post baseline treatment
  Response status at each timepoint of the follow-up period and at 2 years post-treatment. Definitions of responder eyes include:
  1. Eyes whose LogMAR BCVA improves (i.e. decreases) by ≥ 0.3 LogMAR (equivalent to a gain of ≥ 15 ETDRS letters) compared to baseline.
  2. Eyes whose LogMAR BCVA does not increase (i.e. worsen) by ≥ 0.3 LogMAR (equivalent to eyes that lose ≤ 15 ETDRS letters) compared to baseline.
  3. Eyes whose LogMAR visual acuity is < 1.0 (i.e. better than LogMAR 1.0, equivalent to better than Snellen acuity of 20/200).
Spectral-Domain - Optical Coherence Tomography (SD-OCT) parameter | at 1.5-Year and 2-Years post baseline treatment
  Parameters measured with SD-OCT over time and at 1.5 and 2-years post baseline treatment. The change from baseline will be the response. Analysis will be performed mainly for second affected/not yet affected eyes treated with GS010 versus placebo and also for first affected eyes receiving GS010 as well
Humphrey Visual Field (HVF) parameter | at 1.5-Year and 2-Years post baseline treatment
  Parameters measured with HVF 30-2 over time and at 1.5 and 2-years post baseline treatment. The change from baseline will be the response. Analysis will be performed mainly for second affected/not yet affected eyes treated with GS010 versus placebo and also for first affected eyes receiving GS010 as well
Pelli Robson Low Vision Contrast Sensitivity parameter | at 1.5-Year and 2-Years post baseline treatment
  Parameters measured with Pelli Robson Low Vision Contrast Sensitivity over time and at 1.5 and 2-years post baseline treatment. The change from baseline will be the response. Analysis will be performed mainly for second affected/not yet affected eyes treated with GS010 versus placebo and also for first affected eyes receiving GS010 as well
Quality of Life: Visual Functioning Questionnaire-25 | at 1.5-Year and 2-Years post baseline treatment
  Visual Functioning Questionnaire-25 at 1.5 and 2-years post-treatment
Quality of Life: 36-Item Short Form Health Survey, version 2 Questionnaire | at 1.5-Year and 2-Years post baseline treatment
  36-Item Short Form Health Survey, version 2 Questionnaire at 1 and 2-years post-treatment.

OTHER OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) | up to 2-Years post baseline treatment
  Adverse events (AEs) and serious adverse events (SAEs), including those that are treatment-emergent and non-treatment-emergent, throughout the study period and at each study visit. Incidence and severity of systemic and local (ocular) AEs and SAEs will be determined at each clinical site and for the entire study cohort.
Physical examinations | At 2-Years post baseline treatment
  Results of physical examinations
Electrocardiograms | At 2-Years post baseline treatment
  Results of Electrocardiograms (ECGs)
Laboratory results | At 2-Years post baseline treatment
  Results of laboratory tests from blood collection
Immune response evaluations | Up to 2-Years post baseline treatment
  Results of immune response evaluations
  1. Time course of the humoral immune response measured with Neutralizing Antibodies (Nab) against Adeno-associated virus vector 2 (AAV2)
  2. Time course of the cellular immune response against AAV2
Blood Bio-dissemination of AAV2 Vector DNA | up to 4 weeks post-treatment
  Results of bio-dissemination testing up to 4-weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Newman, MD, Principal Investigator — Emory University Hospital Atlanta, Georgia, United States, 30322
Locations (13):
- United States (7):
  - Doheny Eye Center UCLA Pasadena, Pasadena, California
  - University of Colorado Health Eye Center, Aurora, Colorado
  - Emory Healthcare - The Emory Clinic, Atlanta, Georgia
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wills Eye Institute - Ocular Oncology Service, Philadelphia, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
- Universitair Ziekenhuis Gent, Ghent, Belgium
- CHNO Les Quinze Vingts, Paris, France
- IRCCS Istituto delle Scienze Neurologiche di Bologna UOC Clinica Neurologica, Bologna, Italy
- Hospital Universitario Ramon y Cajal, Madrid, Spain
- Taipei Veterans General Hospital, Taipei, Taiwan
- Moorfields Eye Hospital, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Carelli V, Newman NJ, Yu-Wai-Man P, Biousse V, Moster ML, Subramanian PS, Vignal-Clermont C, Wang AG, Donahue SP, Leroy BP, Sergott RC, Klopstock T, Sadun AA, Rebolleda Fernandez G, Chwalisz BK, Banik R, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA; the LHON Study Group. Indirect Comparison of Lenadogene Nolparvovec Gene Therapy Versus Natural History in Patients with Leber Hereditary Optic Neuropathy Carrying the m.11778G>A MT-ND4 Mutation. Ophthalmol Ther. 2023 Feb;12(1):401-429. doi: 10.1007/s40123-022-00611-x. Epub 2022 Nov 30. PMID 36449262
- See also: GenSight Biologics website — http://www.gensight-biologics.com